CLINICAL TRIAL: NCT03011658
Title: Assessment of Anxiety and Depression in Symptomatic Oral Lichen Planus
Brief Title: Serum Cortisol Levels in Patients With Anxiety and Depression With Symptomatic Oral Lichen Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, NALLAN CHAITANYA, Principal investigator, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PMVIDS&RC/IEC/OMR/DN/0004-15
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Oral Lichen Planus Related Stress
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GROUP A (Placebo Comparator): 5 ml of venous blood will be obtained from this group who do not have oral lichen planus and suffering from anxiety and/or depression. They will be administered a HADS standard questionnaire and their stress related issues calculated accordingly. This group has 30 patients totally
  Interventions: Procedure: venepuncture
- GROUP B (Other): The group has 30 oral symptomatic lichen planus diagnosed patients also suffering with anxiety and/or depression. 5 ml of venous blood will be obtained from them for serum cortisol level analysis. HADS questionnaire will be administered for this group for evaluation of levels of anxiety and depression
  Interventions: Procedure: venepuncture

INTERVENTIONS:
Procedure: venepuncture — for both the groups, HADS questionnaire will be administered to assess the levels of anxiety and depression. The placebo group ( group A) will not be having subjects suffering from oral lichen planus

SUMMARY:
Oral lichen planus (OLP) is a T-cell mediated chronic immunological disease directed to a still unknown antigen. It is a mucocutaneous and a psychosomatic disorder, with unknown prevalence rate; however studies suggest an incidence of 0.02 to 0.22% among the Indian population. 75% of patients with cutaneous lichen planus also experience oral lesions and may be precipitated or exacerbated by psychosocial stressors.

In conditions like pain, anxiety and stress, many metabolic and endocrine changes occur in the body, the most common effect of which is increased cortisol level in blood. This hormone is a 21-carbon corticosteroid secreted by adrenal cortex and regulates the metabolism of carbohydrates, fats, proteins and water. Also known as stress hormone, cortisol is a decisive index in stressful situations.

This study is intended to correlate the serum cortisol levels with anxiety and depression in patients with symptomatic oral lichen planus. This study attempts to evaluate psychological anxiety and depression in oral lichen planus subjects using Hospital Anxiety and Depression Scale ( HADS) and correlating with their serum cortisol levels.

To understand and explore the etiopathogenesis for better management of oral lichen planus.

DETAILED DESCRIPTION:
Oral lichen planus (OLP) is a T-cell mediated chronic immunological disease directed to a still unknown antigen. It is a mucocutaneous and a psychosomatic disorder, with unknown prevalence rate; however studies suggest an incidence of 0.02 to 0.22% among the Indian population. 75% of patients with cutaneous lichen planus also experience oral lesions and may be precipitated or exacerbated by psychosocial stressors.

In conditions like pain, anxiety and stress, many metabolic and endocrine changes occur in the body, the most common effect of which is increased cortisol level in blood. This hormone is a 21-carbon corticosteroid secreted by adrenal cortex and regulates the metabolism of carbohydrates, fats, proteins and water. Also known as stress hormone, cortisol is a decisive index in stressful situations.

This study is intended to correlate the serum cortisol levels with anxiety and depression in patients with symptomatic oral lichen planus.

ELIGIBILITY:
Inclusion criteria

* Clinical features with burning sensation on eating spicy food.
* Patients with symptomatic Oral lichen planus evaluated clinically and histologically.

Exclusion criteria:

* Patients not willing to be part of the study.
* Patients who are on corticosteroid therapy.
* Patients with endocrinal disorders which can alter adrenal gland function.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Serum- cortisol levels from venous blood. | 1 year

SECONDARY OUTCOMES:
Hospital Anxiety and Depression scale | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: NALLAN chaitanya, MDS, Principal Investigator — READER
Locations (1):
- Panineeya Institute of Dental Sciences, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No